CLINICAL TRIAL: NCT04155580
Title: A Phase 1, Parallel, Open-Label Study of the Safety and Tolerability, Pharmacokinetics, and Antileukemic Activity of ASTX660 as a Single Agent and in Combination With ASTX727 in Subjects With Relapsed/Refractory (R/R) Acute Myeloid Leukemia (AML)
Brief Title: A Study of ASTX660 as a Single Agent and in Combination With ASTX727 in Subjects With Relapsed/Refractory Acute Myeloid Leukemia (AML)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study halted prematurely and will not resume; participants are no longer being examined or receiving intervention
Sponsor: Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ASTX660-02
Record Dates: First submitted 2019-11-05; First posted 2019-11-07 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; Bone marrow; CMML; MDS; ASTX727; ASTX660; cIAP1; Cellular inhibitor of apoptosis protein; XIAP; CDAi; Cytidine deaminase inhibitor; Cedazuridine; Decitabine; Acute myeloid leukemia; Chronic myelomonocytic leukemia; Myelodysplastic syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes | interventions — ASTX-660; decitabine and cedazuridine drug combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1 (Experimental): ASTX660 once daily (Days 1-7 and 15-21 per 28-day cycle) + ASTX727 FDC once daily (Days 1-5 per 28-day cycle)
  Interventions: Drug: ASTX660; Drug: ASTX727
- Part 2 (Experimental): ASTX660 once daily (Days 1-7 and 15-21 per 28-day cycle) as a single agent or in combination with ASTX727 FDC once daily (Days 1-5 per 28-day cycle)
  Interventions: Drug: ASTX660; Drug: ASTX727
- Part 3 (Experimental): ASTX660 at the recommended dose for expansion identified in Part 2 + ASTX727 FDC once daily (Days 1-5 per 28-day cycle)
  Interventions: Drug: ASTX660; Drug: ASTX727

INTERVENTIONS:
Drug: ASTX660 — Capsule for oral administration
Drug: ASTX727 — Tablet for oral administration
  Other Names: cedazuridine + decitabine

SUMMARY:
To evaluate the safety, pharmacokinetics (PK), and efficacy of ASTX660 when given alone and in combination with ASTX727 in participants with relapsed/refractory (R/R) acute myeloid leukemia (AML). The duration of the study is expected to be approximately 30 months.

DETAILED DESCRIPTION:
This is a three-part dose escalation and dose expansion Phase 1 study of ASTX660 alone and in combination with ASTX727 in adults with R/R AML.

Part 1 is an open-label, single arm, dose escalation with ASTX660 in combination with ASTX727 at the standard fixed dose combination (FDC).

Part 2 is an open-label, randomized, dose escalation intended to evaluate ASTX660 as a monotherapy and ASTX660 in combination with ASTX727 FDC.

Part 3 is an exploratory single arm dose expansion to further expand the number of participants treated with ASTX660 in combination with ASTX727 FDC.

ELIGIBILITY:
Inclusion Criteria:

1. Have a projected life expectancy of at least 12 weeks, as assessed by the Investigator.
2. Have histological confirmation of AML by World Health Organization (WHO) 2016 criteria and are either:

   1. refractory to intensive induction chemotherapy OR
   2. relapsed after intensive induction chemotherapy or stem cell transplant OR
   3. relapsed after or refractory to treatment with molecularly targeted and/or low-intensity chemotherapeutic regimens.
3. Have an Eastern Cooperative Oncology Group (ECOG) Performance status of 0 to 2.
4. Have adequate renal function as demonstrated by measured or calculated creatinine clearance ≥60 mL/min.
5. Have adequate liver function as demonstrated by:

   1. Aspartate aminotransferase (AST) ≤2.5 × upper limit of normal (ULN)
   2. Alanine aminotransferase (ALT) ≤2.5 × ULN
   3. Bilirubin ≤1.5 × ULN - unless considered due to leukemic organ involvement.
6. Women of child-bearing potential (according to recommendations of the Clinical Trial Facilitation Group [CTFG]) must not be pregnant or breastfeeding and must have a negative pregnancy test at screening.

Exclusion Criteria:

1. Poor medical risk in the investigator's opinion because of systemic diseases in addition to the cancer under study, for example, uncontrolled infections.
2. Known clinically active central nervous system (CNS) leukemia.
3. BCR-ABL-positive leukemia (chronic myelogenous leukemia in blast crisis).
4. Diagnosis of acute promyelocytic leukemia (M3 AML or APML).
5. Second malignancy currently requiring active therapy, except breast or prostate cancer stable on or responding to endocrine therapy.
6. Graft Versus Host Disease (GVHD), or any GVHD requiring treatment with immunosuppression. Any GVHD treatment (including calcineurin inhibitors) must be discontinued at least 28 days prior to Day 1 of study treatment.
7. Presence of persistent toxicities of Grade >1 from prior treatment including chemotherapy, targeted therapy, immunotherapy, experimental agents, radiation, and surgery (except for alopecia).
8. Hypersensitivity to decitabine, ASTX727, ASTX660, or any of their excipients.
9. Liver cirrhosis, or chronic liver disease Child-Pugh Class B or C.
10. Life-threatening illness, significant organ system dysfunction, or other condition that, in the investigator's opinion, could compromise participant safety, or the integrity of study outcomes, or interfere with the absorption or metabolism of ASTX660 or ASTX727.
11. History of, or at risk for, cardiac disease.
12. Known human immunodeficiency virus (HIV), active hepatitis B virus (HBV), or active hepatitis C virus (HCV) infection (participants with laboratory evidence of no active replication will be permitted).
13. Known significant mental illness or other conditions, such as active alcohol or other substance abuse that, in the opinion of the investigator, predispose the participant to high risk of noncompliance with the protocol treatment or assessments.
14. Treated with any investigational therapy within 2 weeks of the first dose of study treatment or treatment with a myelosuppressive therapy within 4 weeks of the first dose of study treatment.
15. In Parts 1 and 2, prior treatment with decitabine for more than 2 cycles. In Part 3, any treatment with an HMA (azacitidine or decitabine, for more than one cycle).
16. Inability to swallow oral medication or inability or unwillingness to comply with the administration requirements related to ASTX660-02 (Note: G-tube administration is not allowed).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-01-14 (Actual)

PRIMARY OUTCOMES:
Safety Assessment: Number of participants with treatment-emergent adverse events (TEAEs) | Up to 30 months

SECONDARY OUTCOMES:
Response rate: Number of participants achieving complete response (CR), complete response with incomplete hematological recovery (CRi), and partial response (PR) as determined by the European LeukemiaNet (ELN) 2017 response criteria for AML | Up to 30 months
Time to response: Time from first dose to the first documented evidence of response | Up to 30 months
Duration of response: Time from the start of response until disease progression or relapse | Up to 30 months
Overall survival: Time since first dose until death due to any cause | Up to 30 months
Composite complete response: Number of participants (sum of CR+CRi) | Up to 30 months
Complete response with partial hematological recovery (CRh): Number of participants | Up to Month 30
Pharmacokinetic parameter: Area under the curve (AUC) | On Days 1, 5 and 6 of Cycle 1 and Day 1 of Cycle 2 (28 days per cycle)
Pharmacokinetic parameter: Maximum plasma concentration (Cmax) | On Days 1, 5 and 6 of Cycle 1 and Day 1 of Cycle 2 (28 days per cycle)
Pharmacokinetic parameter: Minimum plasma concentration (Cmin) | On Days 1, 5 and 6 of Cycle 1 and Day 1 of Cycle 2 (28 days per cycle)
Pharmacokinetic parameter: Time to reach maximum plasma concentration (Tmax) | On Days 1, 5 and 6 of Cycle 1 and Day 1 of Cycle 2 (28 days per cycle)
Pharmacokinetic parameter: Half-life (t½) | On Days 1, 5 and 6 of Cycle 1 and Day 1 of Cycle 2 (28 days per cycle)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - University of California San Francisco, San Francisco, California
  - Smilow Cancer Hospital, New Haven, Connecticut
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Northside Hospital - The Blood and Marrow Transplant Group of Georgia, Atlanta, Georgia
  - The University of Chicago Medical Center, Chicago, Illinois
  - Franciscan Health Indianapolis (Blood and Marrow Transplantation), Indianapolis, Indiana
  - The University of Kansas Clinical Research Center, Fairway, Kansas
  - Mayo Clinic, Rochester, Minnesota
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - New York University Langone Health, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Vanderbilt - Ingram Cancer Center, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No